CLINICAL TRIAL: NCT02024542
Title: Genetic and Biochemical Characteristics of Medically-Complicated Obesity and Response to Bariatric Surgery
Brief Title: Metabolic Responses to Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 228969
Record Dates: First submitted 2013-12-25; First posted 2013-12-31 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Morbid Obesity
Keywords: Bariatric Surgery; Obesity; Metabolic syndrome; Diabetes; Liver Disease
MeSH Terms: conditions — Obesity, Morbid; Obesity; Metabolic Syndrome; Diabetes Mellitus; Liver Diseases | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, feces, liver, adipose tissue, GI tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Weight Loss Surgery - Healthy: Patients consented to participate have met the NIH criteria for Bariatric Surgery and have completed the normal pre-operative work up including nutritional counseling, psychological evaluation, and all necessary studies to rule out other co-morbid conditions prior to surgery. Patients do not have metabolic syndrome.
  Interventions: Other: Surgery
- Weight Loss Surgery - Metabolic Syndrome: Patients consented to participate have met the NIH criteria for Bariatric Surgery and have completed the normal pre-operative work up including nutritional counseling, psychological evaluation, and all necessary studies to rule out other co-morbid conditions prior to surgery. Patients have metabolic syndrome.
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery — Patients wishing to participate in the research will complete all necessary pre-operative work-up labs, testing & counseling, complete and sign the informed consent. During weight loss surgery a small amount of subcutaneous and omental fat will be collected for analysis, with subsequent blood collection post surgery for analysis.

SUMMARY:
Research the genetic and biomechanical markers of human adipose tissue on patients with morbid obesity. Additional tissue/fluid collection is also gathered during the time of surgery.

DETAILED DESCRIPTION:
Study participation by invitation after complete pre-surgical work up at UC Davis Health System. Patients will be invited to participate if they meet all inclusion criteria's after completing all necessary clinical visits including lab studies, counseling, and participation in educational programs. During the pre-operative visit patients interested in participation will complete all necessary consent documentation. Pre-operative labs (blood and urine) will be collected along with additional blood, urine, and fecal samples will be collected pre-operatively. During surgery (Roux-en-Y Gastric Bypass surgeries only) tissue collection will include subcutaneous & omental fat, jejunum, and liver biopsy. Post surgery patient will be observed for weight loss and resolution of co-morbidities. At designated times post surgery when lab studies are ordered additional blood/urine samples will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Meet NIH Criteria for Bariatric Surgery
* Between the Age of 18-55
* Dyslipidemia controlled with medication
* Impaired glucose metabolism or type 2 diabetes

Exclusion Criteria:

* Uncontrolled Metabolic syndrome (uncontrolled diabetes, htn, dyslipidemia), one or all conditions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients only (currently).
Study Population: Patients who present for bariatric surgery to treat morbid obesity.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-02; Primary Completion 2035-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Tensile Strength of White Adipose Tissue | July 2012
  During the research tissue samples were compared between healthy obese patients (no diabetes, controlled HTN, no dyslipidemia) with tissue samples collected on non-healthy obese patients (type II diabetes) and using fat collected from mice as a control.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R Ali, MD, Principal Investigator — University of California Davis Health System
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/studying-metabolic-responses-to-bariatric-surgery-425960/